CLINICAL TRIAL: NCT04691037
Title: Improving the Clinical Management of Stable Chest Pain Based on Imaging: a Registry of Computed Tomography Coronary Angiography
Brief Title: CCTA Improves Clinical Management of Stable Chest Pain
Acronym: CICM-SCP
Status: Recruiting | Type: Observational
Sponsor: Tianjin Chest Hospital (Other)
Responsible Party: Principal Investigator, Zhou Jia, Doctor, Tianjin Chest Hospital
Other Study IDs: 2017-KY-004
Record Dates: First submitted 2020-12-29; First posted 2020-12-31 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Coronary Computed Tomography Angiography; Stable Chest Pain; Optimal Medical Therapy; Invasive Coronary Angiography; Revascularization; Major Adverse Cardiovascular Events; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CCTA
  Interventions: Diagnostic Test: CCTA

INTERVENTIONS:
Diagnostic Test: CCTA — All patients underwent CCTA according to established guidelines and local institutional protocols. The imaging data were evaluated using different image post-processing software to comprehensively analyse anatomical, functional and histological information of coronary.

SUMMARY:
The investigator aims to prospectively enroll patients who were referred for coronary computed tomography angiography (CCTA) for the assessment of stable chest pain (SCP) suspected of obstructive coronary artery disease (CAD). All patients underwent CCTA according to established guidelines and local institutional protocols. The imaging data were evaluated using different image post-processing software to comprehensively analyse anatomical, functional and histological information of coronary. This study will determine if CCTA-based imaging evaluation can provide more informaton to improve clinical management for SCP, including fewer MACE and better decision-making of downstream investigations and therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic patients with SCP suspected of obstructive CAD.
* referred for CCTA for the assessment of SCP.
* ≥18 years of age.
* signed informed consent.

Exclusion Criteria:

* acute coronary syndromes
* previous CAD or coronary revascularization
* nonsinus rhythm
* cardiomyopathy, valvular disease, congenital heart disease or left cardiac insufficiency because of other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were referred for CCTA for the assessment of SCP suspected of CAD.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | 10 years
  Cardiac death and myocardial infarction

SECONDARY OUTCOMES:
Invasive coronary angiography | 10 years
  Invasive coronary angiography occurred at follow-up after CCTA, attributed to CCTA results or unplanned.
Medication prescription | 10 years
  Change for medication prescription of antiplatelet agents, anti-ischemic drugs, lipid-lowering agents, angiotensin-converting enzyme inhibition and so on, attributed to CCTA results or unplanned,
Coronary revascularization | 10 years
  PTCA, PCI or CABG occurred at follow-up after CCTA, attributed to CCTA results or unplanned.
Number of Participants with Death | 10 years
Number of Participants with Stroke | 3 years
Number of Participants with Cardiac death | 10 years
Number of Participants with Myocardial infarction | 10 years

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Beijing Chaoyang Hospital, Beijing, Beijing Municipality
  - Hebei Petrochina Central Hospital, Langfang, Hebei
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - Tianjin First Central Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tan Y, Liu C, Chen T, Li Y, Wang C, Zhao J, Zhou J. Coronary Artery Calcium Score-Weighted Clinical Likelihood Model Performance in Patients with Stable Chest Pain and Coronary Artery Calcium Scores of Zero. Rev Cardiovasc Med. 2024 Mar 4;25(3):85. doi: 10.31083/j.rcm2503085. eCollection 2024 Mar. PMID 39076944
- [Derived] Zhou J, Li C, Zhang H, Liu C, Yang J, Zhao J, Hou Y, Tan Y, Wang H, Li Y, Xie C, Wang M, Wang C, Zhang E, Wang S, Zhao P, Shan D, Liang S, Gao Y, Huo Y, Cong H, Guo Z, Chen Y. Association between Coronary Artery Disease Reporting and Data System-recommended Post-Coronary CT Angiography Management and Clinical Outcomes in Patients with Stable Chest Pain from a Chinese Registry. Radiology. 2023 Jun;307(5):e222965. doi: 10.1148/radiol.222965. PMID 37310243
- [Derived] Jiang H, Feng J, Feng C, Ren P, Ren K, Jin Y, Zhou J. Validation and Comparison of PROMISE and CONFIRM Model to Predict High-Risk Coronary Artery Disease in Symptomatic and Diabetes Mellitus Patients. Rev Cardiovasc Med. 2022 Mar 1;23(3):80. doi: 10.31083/j.rcm2303080. PMID 35345247